CLINICAL TRIAL: NCT03715296
Title: Lenalidomide Based Immunotherapy Efficacy Related Molecular Biomarker in Diffuse Large B-cell Lymphoma
Brief Title: Lenalidomide Based Immunotherapy in the Treatment of DLBCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Other Study IDs: NHL-007
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lenalidomide 25mg — Lenalidomide 25mg/d PO d1-10 Plus Rituximab 375 mg/m2 IV d1, Cyclophosphamide 750mg/m2 IV d2, Doxorubicin 50mg/m2 IV d2, Vincristine 1.4 mg/m2 IV d2, Prednisone 60 mg/m2 PO d2-6 OR Ifosfamide 1500mg/m2/d iv d1-3, Carboplatin 5*[GFR(ml/min)+25]mg/d iv d2, Etoposide 100mg/m2/d iv d1-3,

SUMMARY:
This study is to evaluate the efficacy related molecular biomarker of Lenalidomide plus RCHOP or RICE in the treatment of de novo or Refractory and Relapsed DLBCL patients

ELIGIBILITY:
Inclusion Criteria:

Histologically diagnosed as diffuse large b-cell lymphoma and may provide a desirable lymph node tissue sample (10 paraffin sections or rolls) or lymph node biopsy sample (15 paraffin sections or rolls)

Previously treated with Lenalidomide plus RCHOP regimen in de novo DLBCL or Lenalidomide plus RICE regimen in relapse refractory DLBCL.

No history of stem cell transplantation.

Written informed consent.

Exclusion Criteria:

Chemotherapy or large field radiotherapy within 3 weeks prior to entering the study.

Clinically significant active infection.

Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule.

Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.

Subject has ≥grade 2 peripheral neuropathy or grade 1 with pain within 14 days before enrollment.

Patients who are pregnant or breast-feeding.

HIV infection.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: De novo DLBCL patients / Relapse Refractory DLBCL patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 12 weeks

SECONDARY OUTCOMES:
Progression free survival rate | 1 year
Overall survival rate | 1 year
Overall response rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China